CLINICAL TRIAL: NCT04066361
Title: OPTimizing Treatment Focused Genetic Testing IN Cancer - OPT-IN
Brief Title: OPTimizing Treatment Focused Genetic Testing IN Cancer
Acronym: OPT-IN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Huma Rana, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-068
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer
Keywords: Other Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot (Experimental): * Participant is given a pamphlet introducing genetic testing
  * Participant is given information utilized for clinical, standard of care testing.
  * Will receive genetic information with a virtual interactive Chatbot prior to genetic testing. After the Chatbot education, participant is asked if they would like to proceed with genetic testing.
  * Participant is asked to complete an electronic family history tool
  Interventions: Other: Chatbot
- Video Education (Experimental): * Participant is given a pamphlet introducing genetic testing
  * Participant is given information utilized for clinical, standard of care testing.
  * Participant will watch a brief educational video that is approximately 8 minutes in length about the genetic testing process and what to expect prior to genetic testing. After the video education, participant is asked if they would like to proceed with genetic testing.
  * Participant is asked to complete an electronic family history tool
  Interventions: Other: Video Education

INTERVENTIONS:
Other: Chatbot — Interactive text chat designed to mirror the educational components of a traditional genetic counseling visit
  Arms: Chatbot
Other: Video Education — Brief video designed to mirror the educational components of a traditional genetic counseling visit
  Arms: Video Education

SUMMARY:
This two-part randomized controlled trial aims to evaluate the impact of pre-test video education as compared to pre-test Chatbot education.

DETAILED DESCRIPTION:
In this research study, the investigators are introducing the option of two alternatives to genetic counseling before genetic testing: Chatbot and video education.

The first part of this research study is a Pilot Study, which is the first-time investigators are examining the use of a Chatbot to deliver pre-genetic test education. The Chatbot will converse with you about germline genetic testing by text message.

The Pilot study will enroll 200 participants with a metastatic breast or ovarian cancer diagnosis and will assess the uptake of genetic testing among the two possible groups of pre-genetic test counseling.

The second part of this research study will utilize findings from the Pilot Study for 1000 participants with a diagnosis of breast, ovarian, pancreatic or prostate cancer.

In both parts of this research study, participants will be randomized to either the video education or Chatbot. Participants may request in-person genetic counseling after their respective education prior to testing.

Other studies at both DFCI and outside institutions have started to investigate alternative methods of educating patients about genetic testing. These studies have suggested that alternatives to standard genetic counseling may increase access to genetic testing with similar satisfaction to standard of care.

The investigators are hoping to get a sense of participants' preferences for pre genetic test education, understanding, and reactions to the alternative methods of genetic counseling. The investigators are also hoping to understand preferences for communication of their result and whether any treatment changes have been made after they receive their result.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18
* With a diagnosis of advanced cancer (defined as Stage 3 or 4), or
* Any stage for pancreatic cancer and
* No prior cancer genetic panel testing

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women (if known at the time of participation)
* Prisoners
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The measurement of genetic testing uptake | 2 years
  The proportion of participants who consent to genetic testing in each study arm
Meaningful cancer treatment changes | 2 years
  Assessed by chart review. Participants with positive genetic test results will be reviewed for changes in cancer treatment.
Satisfaction with pre-genetic test education | at time of post-counseling/video pre-result disclosure, on average 3 weeks
  A validated survey of participants' satisfaction with the genetic counseling and testing process will be used. For the survey at the time of post-counseling, the survey for the video education arm consists of 8 questions and the genetic counseling arm contains an additional question about perceived length of the visit. The parameters for measurement are "disagree strongly", "disagree", "neither agree or disagree", "agree", and "agree strongly".

SECONDARY OUTCOMES:
Communication of results with family members | 4 months post-result disclosure
  For those participants who have tested positive for a mutation, 5 items will be asked pertaining to disclosure of genetic testing results to relatives that are derived from previous literature.
Intent to disclose genetic test results | 1 day (at time of intervention)
  Three items will assess participants' intentions to disclose genetic testing results
Cascade testing of family members | 6 month post-result disclosure
  This will evaluate participant's discussions about genetic testing within the family for an understanding of how genetic testing information was communicated
Decisional regret | 4 months post-result disclosure
  5 items will be asked pertaining to reflecting on the decision of the participant about getting genetic testing after learning about their result.
Knowledge of multi-gene panel testing | 1 day (at the time of intervention)
  A 6 item survey evaluating participant's understanding of inherited genetic risk

CONTACTS AND LOCATIONS:
Overall Officials: Huma Q Rana, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: http://innovation@dfci.harvard.edu